CLINICAL TRIAL: NCT01673256
Title: DEtermining Accuracy and TrEnding CharacTerization of AF
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: DETECT AF
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Results first posted 2015-03-18 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SJM Confirm ICM Observational Group
  Interventions: Device: SJM Confirm ICM

INTERVENTIONS:
Device: SJM Confirm ICM

SUMMARY:
The objective of this study is to assess the atrial fibrillation (AF) episode detection when using the SJM(St. Jude Medical) Confirm ICM (Implantable Cardiac Monitor).

ELIGIBILITY:
Inclusion Criteria:

* The subject has been implanted with a SJM Confirm ICM, DM2102.
* The subject has or is suspected to have paroxysmal AF.
* The subject is ≥ 18 years of age.
* The subject is willing and able to provide written Informed Consent (prior to any investigational related procedure).

Exclusion Criteria:

* The subject has persistent (>7 days and ≤1 year or requiring cardioversion), longstanding persistent (continuous AF >1 year) or permanent AF (not attempting to restore sinus rhythm).
* The subject has AF of reversible etiology (e.g. electrolyte imbalance, thyroid disease).
* The subject has a contraindication to Holter recording.
* The subject has already received an active implantable medical device other than the SJM Confirm ICM, DM2102.
* The subject is unable to comply with the follow up schedule.
* The subject is participating in another investigational device or drug investigation.
* The subject is pregnant or is planning to become pregnant during the duration of the investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Lewalter, MD, Principal Investigator — Isar Heart Center Munich
Locations (13):
- Germany (11):
  - Rhön-Klinikum, Herz- und Gefäß-Klinik, Bad Neustadt an der Saale
  - Herz -und Diabeteszentrum, Bad Oeynhausen
  - Charite, Campus Virchow-Klinikum, Berlin
  - Klinikum Coburg, Coburg
  - University of Dresden - Heart Center, Dresden
  - Klinikum Frankfurt Höchst GmbH, Frankfurt
  - Klinikum Ingolstadt GmbH, Ingolstadt
  - Herzzentrum Leipzig, Leipzig
  - Isar Heart Center, Munich
  - Hegau-Bodensee-Kliniken, Singen
  - Schwarzwald-Baar Klinikum GmbH, Villingen-Schwenningen
- Netherlands (2):
  - Albert Schweitzer Hospital, Dordrecht
  - Hagahospital, The Hague

RESULTS

PARTICIPANT FLOW:
Groups:
- SJM Confirm ICM Observational Group: SJM Confirm ICM
Period: Overall Study
Arm/Group | SJM Confirm ICM Observational Group
Started | 90
Completed | 90
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SJM Confirm ICM Observational Group
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 55
Region of Enrollment [Number; unit: participants]
  Netherlands | 5
  Germany | 85
Weight [Mean (Standard Deviation); unit: kg] | 82.4 (16.4)

OUTCOME MEASURES:

1. Primary Outcome: Assess SJM (St. Jude Medical) Confirm ICM (Implantable Cardiac Monitor) Sensitivity and Positive Predictive Values of AF Episodes of at Least 2 Minutes in Length, Utilizing the Data Collected During the Holter Recording.
Description: Sensitivity measures the percentage of the actual duration of AF identified by the Holter monitor (for all AF detections that are ≥2 minutes in duration observed in the study) which are correctly identified as AF by the SJM Confirm ICM.
  Positive Predictive Value measures the percentage of the duration of AF detected (for all AF detections that are ≥2 minutes in duration observed in the study) by the SJM Confirm that is identified as AF by the Holter monitor.
Time Frame: 4 days after Holter starts
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | SJM Confirm ICM Observational Group
Number analyzed (Participants) | 79
percentage
  Duration Sensitivity | 83.9 [71.6 to 96.1]
  Duration Positive Predictive Value | 97.3 [91.9 to 100]

ADVERSE EVENTS:
Arm/Group | SJM Confirm ICM Observational Group
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less